CLINICAL TRIAL: NCT03256513
Title: The Safety and Efficacy of Peri-procedure Blood Pressure Management of Revascularization for Ischemic Cerebral Vascular Disease
Brief Title: The Safety and Efficacy of Peri-procedure Blood Pressure Management of Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University Third Hospital (Other); The 306 Hospital of People's Liberation Army (Other)
Responsible Party: Principal Investigator, lingfeng, clinical investigator, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D161100003816002
Record Dates: First submitted 2017-06-01; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cerebral Revascularization; Ischemic Cerebrovascular Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- model controlling (Experimental): an statistical model for periprocedural blood pressure control
  Interventions: Other: model controlling
- conventional controlling (Active Comparator): an conventional strategy for periprocedural blood pressure control
  Interventions: Other: conventional controlling

INTERVENTIONS:
Other: model controlling — control blood pressure by statistical l model with anticipate lowest peri-procedure risk
  Arms: model controlling
Other: conventional controlling — control blood pressure by conventional strategy
  Arms: conventional controlling

SUMMARY:
Objective: Referring The relation between CEA(Carotid endarterectomy) postoperative blood flow monitoring and blood pressure, and combining patient demographics and preoperative risk factors to establish an applicable individual blood pressure controlling model. By comparing with routine antihypertensive strategies through prospective randomized controlled trials , to provide the best perioperative blood pressure control standards and strategies for each patient ,thus better ensuring the safety and efficacy of CEA .

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patient with carotid artery stenosis>=50% or asymptomatic patient with carotid artery stenosis>=70%, according to DSA or CTA;
* without massive cerebral infarction(infarction area >1/2 territory of middle cerebral artery) confirmed by CT or MRI;
* informed consent acquired.

Exclusion Criteria:

* lesion beyond range limit of procedure (higher than C2);
* target vascular complete occlusion or ipsilateral intracranial artery severe stenosis or complete occlusion cannot be revascularized via CEA procedure
* nonatherosclerotic carotid stenosis, such as vasculitis, dissection, congenital vascular malformation;
* history of instable angina pectoris, myocardial infarction or congestive heart failure within 6 months unable to accept systematic anesthesia;
* history of severe injury, surgery or radiotherapy on neck;
* with comorbid hemorrhagic cerebral disease such as intracranial aneurysm or vascular malformation;
* with comorbid blood system disease causing refractory coagulation dysfunction or rejection to blood or blood products perfusion;
* with other comorbidity, expected life < 2 years;
* severe diabetes mellitus difficult to control, blood sugar >300mg/dl;
* pregnancy or peri-natal period;
* intolerance to systematic anesthesia or surgery after adequate preparation.
* intolerance to peri-procedural drug possible to administrated;
* not cooperating or rejecting to informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2270 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
death | 30 days
  all cause death
ischemic stroke | 30 days
  Ischemic stroke is defined as an acute episode of neurological events with focal symptoms and signs, with a duration of more than 24h and confirmed by imaging.
cardiovascular events | 30 days
  Cardiovascular events were defined as: ECG presentation clearly different from preoperative myocardial ischemia, myocardial infarction, arrhythmia and cardiovascular death.

SECONDARY OUTCOMES:
transient ischemic attack,TIA | 30 days
  transient ischemic attack, TIA is defined as: Patients with new onset of neurological symptoms and / or signs, duration < 24 hours, MRI diffusion weighted imaging (DWI) did not find new infarcts. If MRI DWI showed new lesion, ischemic stroke was defined.
cerebral hemorrhage | 30 days
  cerebral hemorrhage including intracerebral hemorrhage, epidural or subdural hemorrhage, subarachnoid hemorrhage.
hyperperfusion syndrome | 30 days
  Hyperfusion Syndrome is defined as : 30 days after operation, new onset headache, vomiting, mental symptoms, macular edema, focal seizures, neurological dysfunction, or imaging brain edema, visible bleeding, and exception of new ischemic cerebral infarction or other causes.
epilepsy | 30 days
  epilepsy is defined as focal onset, with or without evolution to a bilateral tonic-clonic seizure, confirmed by EEG findings including interictal epileptiform discharges (IEDs), lateralized periodic discharges (LPDs; previously known as periodic lateralized epileptiform discharges [PLEDs]), and generalized periodic discharges (GPDs)

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, Principal Investigator — Department of neurosurgery, Xuanwu hospital
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, China